CLINICAL TRIAL: NCT02933632
Title: Accelerated Rehabilitation Versus Conventional Rehabilitation in Total Hip Arthroplasty: A Randomized Double Blinded Clinical Trial
Brief Title: Accelerated Rehabilitation in Hip Arthroplasty
Acronym: ARTHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Angela Elizabeth Marchisio, Master Degree, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FederalURS
Record Dates: First submitted 2015-04-13; First posted 2016-10-14 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Physiotherapy; Rehabilitation; Clinical Trials; Accelerated rehabilitation; Hip Replacement Arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Assistance Protocol-SAP (Active Comparator): Patients underwent physical therapy once a day. Patients receive intervention by Physical Therapy-SAP.
  Interventions: Other: Physical Therapy-SAP
- Accelerated Rehabilitation Protocol-ARP (Active Comparator): Patients underwent physical therapy three times a day. Patients receive intervention by Physical Therapy-ARP.
  Interventions: Other: Physical Therapy-ARP

INTERVENTIONS:
Other: Physical Therapy-SAP — * Day 1) Patients started approach after discharged anesthesia. Patients received verbal orientation and demonstration of the physiotherapy exercises that would strengthen muscles (gluteal and thigh). They were oriented to the decubitus changes and how to leave bed. They practiced 3 repetitions of 12 complete movements for each exercise;
  * Day 2) Patients repeated the exercises learned from day 1. Following the proposed activities patients received verbal instructions on gait training and then starting gait training. Patients started gait training on this second day only if they felt safe and claimed that their pain was controlled. Otherwise, training was postponed to the next day;
  * Day 3) Patients repeated the day 2. And the patient who had not started gait training in the day 2, began it on the day 3;
  * Day 4 and other days) Patients repeated the gait training until the discharge date.
  Arms: Standard Assistance Protocol-SAP
Other: Physical Therapy-ARP — * Day 1-1°approach) Patients started after discharged anesthesia. Received verbal orientation and demonstration of the physiotherapy exercises that would strengthen muscles (gluteal and thigh). They were oriented to the decubitus changes and how to leave bed. They practiced 3 repetitions of 12 complete movements for each exercise;
  * Day 1-2°approach) Patients repeated the exercises learned from day 1-1°approach. Following patients received verbal instructions on gait training and then starting gait training. Patients started gait training on this Day 1-2°approach only if they felt safe and claimed that their pain was controlled. Otherwise, training was postponed to next approach;
  * Day 1-3°approach) Patients repeat the day 1-2°approach. And the patient, who had not started gait training in the day 1 - second approach, began it in this third approach;
  * Day 2) Patients repeated three times the day 1-3°approach;
  * Day 3) Patients repeated three times the day 1-3°approach.
  Arms: Accelerated Rehabilitation Protocol-ARP

SUMMARY:
Accelerated rehabilitation protocol in Total Hip Arthroplasty (THA-AR).

DETAILED DESCRIPTION:
The accelerated rehabilitation protocol in Total Hip Arthroplasty (THA-AR) was designed to improve the functionality and optimize early discharge of patients undergoing THA surgery. This study compared physical therapy protocol in Total Hip Arthroplasty (THA-PT) already deployed in Porto Alegre Clinical Hospital with THA-AR.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Public Health System of our Country that were admitted with hip osteoarthritis diagnose and submitted to a total hip arthroplasty surgery in the Hospital de Clínicas de Porto Alegre (HCPA).

Exclusion Criteria:

* Patients who refused to participate in this study;
* Patients lived in another city;
* Patients undergoing surgery for total hip arthroplasty due to hip fracture;
* Patients with cognitive disorders or diseases that adversely affect its cognitive function (Alzheimer's disease, senile dementia).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Merle D'Aubigné and Postel score | From the moment of hospitalization until the day of hospital discharge, assessed up to four days.

SECONDARY OUTCOMES:
Length of hospital stay | From the moment of hospitalization until the day of hospital discharge, assessed up to four days.
Muscle strength force | From the moment of hospitalization until the day of hospital discharge, assessed up to four days.
  Measured based on Kendall's criteria. Measured in the operated hip.
Goniometry | From the moment of hospitalization until the day of hospital discharge, assessed up to four days.
  Evaluate the range of motion in flexion, extension, adduction, abduction, and internal and external rotation in the operated hip.
Time to beginning the gait. | From the date of hospitalization until the day that began gait, assessed up to four days.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Galia, Doctor, Principal Investigator — Federal University Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Federal University Rio Grande do Sul, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marchisio AE, Ribeiro TA, Umpierres CSA, GalvAo L, Rosito R, Macedo CAS, Galia CR. Accelerated rehabilitation versus conventional rehabilitation in total hip arthroplasty (ARTHA): a randomized double blinded clinical trial. Rev Col Bras Cir. 2020;47:e20202548. doi: 10.1590/0100-6991e-20202548. Epub 2020 Aug 12. English, Portuguese. PMID 32844909
- See also: Link to publication — https://doi.org/10.1590/0100-6991e-20202548